CLINICAL TRIAL: NCT02522871
Title: International Randomized Trial to Evaluate The Effectiveness of The Portable Organ Care System (OCS™) Liver For Preserving and Assessing Donor Livers for Transplantation (OCS Liver PROTECT Trial)
Brief Title: OCS Liver PROTECT Trial: Preserving and Assessing Donor Livers for Transplantation
Acronym: PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCS-LVR-092014
Record Dates: First submitted 2015-08-11; First posted 2015-08-13 (Estimated); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2022-01

CONDITIONS: Liver Transplantation; Liver Preservation for Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCS Liver System (Experimental): OCS Liver System
  Interventions: Device: OCS™ Liver System
- Control (Other): Standard of care (ice)
  Interventions: Other: Control

INTERVENTIONS:
Device: OCS™ Liver System
  Arms: OCS Liver System
Other: Control
  Arms: Control

SUMMARY:
A prospective, phased-pivotal, international randomized trial to evaluate the effectiveness of the OCS™ Liver to preserve and assess donor livers intended for transplantation.

DETAILED DESCRIPTION:
The OCS™ Liver PROTECT Trial is a two-armed, multicenter, prospective, randomized, controlled pivotal trial to evaluate the effectiveness and safety of the OCS Liver to preserve and assess donor livers intended for transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Registered male or female primary Liver transplant candidate
* Age ≥18 years old
* Signed: 1) written informed consent document and 2) authorization to use and disclose protected health information

Exclusion Criteria:

* Acute, fulminant liver failure
* Prior solid organ or bone marrow transplant
* Chronic use of hemodialysis or diagnosis of chronic renal failure, defined as chronic serum creatinine of >3 mg/dl for >2 weeks and/or requiring hemodialysis
* Multi-organ transplant
* Ventilator dependent
* Dependent on > 1 IV inotrope to maintain hemodynamics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-01-24 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elbetanony, MD, Study Director — TransMedics
Locations (20):
- United States (20):
  - University of California San Diego, La Jolla, California
  - Scripps, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Tampa General, Tampa, Florida
  - Emory, Atlanta, Georgia
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai, New York, New York
  - Montefiore Einstein Center for Transplantation, The Bronx, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Methodist University Hospital, Memphis, Tennessee
  - University of Texas Southwest, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - University of Texas San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Markmann JF, Abouljoud MS, Ghobrial RM, Bhati CS, Pelletier SJ, Lu AD, Ottmann S, Klair T, Eymard C, Roll GR, Magliocca J, Pruett TL, Reyes J, Black SM, Marsh CL, Schnickel G, Kinkhabwala M, Florman SS, Merani S, Demetris AJ, Kimura S, Rizzari M, Saharia A, Levy M, Agarwal A, Cigarroa FG, Eason JD, Syed S, Washburn WK, Parekh J, Moon J, Maskin A, Yeh H, Vagefi PA, MacConmara MP. Impact of Portable Normothermic Blood-Based Machine Perfusion on Outcomes of Liver Transplant: The OCS Liver PROTECT Randomized Clinical Trial. JAMA Surg. 2022 Mar 1;157(3):189-198. doi: 10.1001/jamasurg.2021.6781. PMID 34985503

RESULTS

PARTICIPANT FLOW:
Groups:
- OCS Liver System: Organ Care System (OCS) Liver
- Control: Ischemic cold storage (ICS)
Period: Overall Study
Arm/Group | OCS Liver System | Control
Started (Enrolled and received liver allograft) | 153 | 147
As-Treated and Safety Population | 153 | 146
Modified Intent to Treat Population | 152 | 146
Per Protocol Population | 151 | 142
Completed (Completing the 12 month visit.) | 142 | 133
Not Completed | 11 | 14
Not completed — Protocol Violation | 1 | 4
Not completed — Treated without randomization | 1 | 0
Not completed — Death | 9 | 9
Not completed — Died in operating room prior to transplant | 0 | 1

BASELINE CHARACTERISTICS:
Population: As Treated Population
Groups:
- OCS Liver: Organ Care System (OCS) Liver
- Total: Total of all reporting groups
Arm/Group | OCS Liver | Control | Total
Number analyzed (Participants) | 153 | 146 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.07 (10.332) | 58.59 (10.043) | 57.81 (10.204)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 46 | 97
  Male | 102 | 100 | 202
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 20 | 39
  Not Hispanic or Latino | 123 | 119 | 242
  Unknown or Not Reported | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 8 | 20
  White | 129 | 131 | 260
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 4 | 13
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.67 (5.383) | 29.51 (5.513) | 29.59 (5.438)
Model for End-stage Liver Disease (MELD) Score [Mean (Standard Deviation); unit: scores on a scale] — Model for End-Stage Liver Disease (MELD) score is based on lab results and is provided to patients based on how urgently they need a liver transplant in the next three months. The MELD score can range from 6 (less ill) to 40 (gravely ill).
  scores on a scale | 28.4 (6.90) | 28.0 (5.71) | 28.2 (6.34)
Primary Diagnosis [Count of Participants; unit: Participants]
  Cholestatic diseases | 9 | 8 | 17
  Chronic hepatitis | 27 | 36 | 63
  Alcoholic cirrhosis | 54 | 48 | 102
  Metabolic diseases | 6 | 6 | 12
  Primary hepatic tumors | 14 | 15 | 29
  NASH | 24 | 20 | 44
  Other | 19 | 13 | 32
Donor Age [Mean (Standard Deviation); unit: years] — Population: Donor Liver Population As Treated. Donor Liver Population As Treated consists of all donor livers for which the potential recipient was randomized, and preservation was initiated using OCS or control. However, one donor liver was excluded due to non-randomization, therefore bringing the Donor Liver Population As Treated to 152 from 153.
  years
    number analyzed (Participants) | 152 | 146 | 298
    (all) | 45.84 (14.904) | 46.96 (15.223) | 46.39 (15.046)
Donor age >= 40 years [Count of Participants; unit: Participants] — Population: Donor Liver Population As Treated. Donor Liver Population As Treated consists of all donor livers for which the potential recipient was randomized, and preservation was initiated using OCS or control. However, one donor liver was excluded due to non-randomization, therefore bringing the Donor Liver Population As Treated to 152 from 153.
  Participants
    number analyzed (Participants) | 152 | 146 | 298
    (all) | 102 | 93 | 195
Donor total cross-clamp time >= 6 hours [Count of Participants; unit: Participants] — Population: Donor Liver Population As Treated. Donor Liver Population As Treated consists of all donor livers for which the potential recipient was randomized, and preservation was initiated using OCS or control. However, one donor liver was excluded due to non-randomization, therefore bringing the Donor Liver Population As Treated to 152 from 153.
  Participants
    number analyzed (Participants) | 152 | 146 | 298
    (all) | 48 | 56 | 104
DCD age <=55 years [Count of Participants; unit: Participants] — Population: Donor Liver Population As Treated. Donor Liver Population As Treated consists of all donor livers for which the potential recipient was randomized, and preservation was initiated using OCS or control. However, one donor liver was excluded due to non-randomization, therefore bringing the Donor Liver Population As Treated to 152 from 153.
  Participants
    number analyzed (Participants) | 152 | 146 | 298
    (all) | 28 | 13 | 41
Steatotic liver >0% and <=40% macrosteatosis [Count of Participants; unit: Participants] — Population: Donor Liver Population As Treated. Donor Liver Population As Treated consists of all donor livers for which the potential recipient was randomized, and preservation was initiated using OCS or control. However, one donor liver was excluded due to non-randomization, therefore bringing the Donor Liver Population As Treated to 152 from 153.
  Participants
    number analyzed (Participants) | 152 | 146 | 298
    (all) | 95 | 86 | 181

OUTCOME MEASURES:

1. Primary Outcome: Participants With Early Liver Allograft Dysfunction (EAD)
Description: Participants with Early liver Allograft Dysfunction (EAD) or primary non-function, defined as presence of one or more of the following criteria: AST level > 2000 IU/ml within the first 7 postoperative days; Bilirubin ≥ 10 mg/dl on postoperative day 7; INR ≥ 1.6 on postoperative day 7; or Primary non-functioning graft within the first 7 days (defined as irreversible graft dysfunction requiring emergency liver re-transplantation or death, in the absence of immunologic or surgical causes)
Time Frame: 7 days
Population: 1 subject in each arm (OCS Liver and Control) has missing data and therefore the overall number of participants analyzed is different than the number reported in the Participant Flow.
Measure: Count of Participants; unit: Participants
Groups:
- OCS Liver - Per Protocol: Organ Care System (OCS) Liver - Per protocol population
- Control - Per-protocol: Ischemic cold storage (ICS) - Per-protocol population
- OCS Liver - mITT: Organ Care System (OCS) Liver - mITT population
- Control - mITT: Ischemic cold storage (ICS) - mITT population
Arm/Group | OCS Liver - Per Protocol | Control - Per-protocol | OCS Liver - mITT | Control - mITT
Number analyzed (Participants) | 150 | 141 | 151 | 145
Participants | 27 | 44 | 27 | 47
Statistical Analysis 1: Comparison: OCS Liver - Per Protocol vs Control - Per-protocol; Test type: Non-Inferiority — non-inferiority margin = 0.075; p < 0.0001, one-sided Farrington and Manning; Difference of Proportion = -0.132, 95% CI 1-sided [upper limit -0.049]
Statistical Analysis 2: Comparison: OCS Liver - mITT vs Control - mITT; Test type: Non-Inferiority — non-inferiority margin = 0.075; p < 0.0001, one-sided Farrington and Manning; Difference of Proportion = -0.145, 95% CI 1-sided [upper limit -0.062]

2. Primary Outcome: Primary Safety Endpoint: Liver Graft-related Serious Adverse Events (LGRSAEs) up to 30-days Post-transplant Per Patient
Description: Defined as the average number of LGRSAEs (Liver Graft-Related Serious Adverse Event) up to the 30-day follow-up after transplantation per patient.
Time Frame: 30 days
Population: As Treated Population
Measure: Mean (Standard Deviation); unit: Events per patient
Arm/Group | OCS Liver | Control
Number analyzed (Participants) | 153 | 146
Events per patient | 0.046 (.210) | 0.075 (0.265)
Statistical Analysis 1: Comparison: OCS Liver vs Control; Test type: Non-Inferiority — non-inferiority margin of 1.0; p < 0.0001, t-test, 1 sided; Mean Difference (Final Values) = -0.030, 95% CI 2-sided [-0.084 to 0.025]

3. Secondary Outcome: Patient Survival at Day 30 After Transplant
Description: Patient survival at day 30 after transplantation
Time Frame: 30 days after transplant
Measure: Count of Participants; unit: Participants
Groups:
- OCS Liver - Per-protocol: Organ Care System (OCS) Liver - Per-protocol
- Control - Per-protocol: Ischemic cold storage (ICS) - Per-protocol
- OCS Liver - mITT: Organ Care System (OCS) Liver - mITT
- Control - mITT: Ischemic cold storage (ICS) - mITT
Arm/Group | OCS Liver - Per-protocol | Control - Per-protocol | OCS Liver - mITT | Control - mITT
Number analyzed (Participants) | 151 | 142 | 152 | 146
Participants | 150 | 141 | 151 | 145
Statistical Analysis 1: Comparison: OCS Liver - Per-protocol vs Control - Per-protocol; Test type: Non-Inferiority — non-inferiority margin = 0.075; p = 0.0004, one-sided Farrington and Manning; Difference of Proportion = -0.000, 95% CI 1-sided [upper limit 0.036]
Statistical Analysis 2: Comparison: OCS Liver - mITT vs Control - mITT; Test type: Non-Inferiority — non-inferiority margin = 0.075; p = 0.0004, one-sided Farrington and Manning; Difference of Proportion = -0.000, 95% CI 1-sided [upper limit 0.036]

4. Secondary Outcome: Patient Survival at Initial Hospital Discharge Post Liver Transplant
Description: Patient survival at initial hospital discharge post liver transplantation
Time Frame: at initial hospital discharge post liver transplant, an average of 11 days
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Liver - Per-protocol | Control - Per-protocol | OCS Liver - mITT | Control - mITT
Number analyzed (Participants) | 151 | 142 | 152 | 146
Participants | 149 | 140 | 150 | 144
Statistical Analysis 1: Comparison: OCS Liver - Per-protocol vs Control - Per-protocol; Test type: Non-Inferiority — non-inferiority margin = 0.075; p = 0.0006, one-sided Farrington and Manning; Difference of Proportion = -0.001, 95% CI 1-sided [upper limit 0.038]
Statistical Analysis 2: Comparison: OCS Liver - mITT vs Control - mITT; Test type: Non-Inferiority — non-inferiority margin = 0.075; p = 0.0006, one-sided Farrington and Manning; Difference of Proportion = -0.001, 95% CI 1-sided [upper limit 0.038]

5. Other Pre Specified Outcome: Evidence of Ischemic Biliary Complications Diagnosed at 6 Months
Description: Number and percentage of Participants with Ischemic Biliary Complications from Day of Transplant through 6 Months Follow-up Visit
Time Frame: 6 months post transplant
Population: per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Liver System | Control
Number analyzed (Participants) | 151 | 142
Participants | 2 | 12

6. Other Pre Specified Outcome: Evidence of Ischemic Biliary Complications Diagnosed at 12 Months
Description: Number and percentage of Participants with Ischemic Biliary Complications from Day of Transplant through 12 Months Follow-up Visit
Time Frame: 12 months post transplant
Population: per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Liver System | Control
Number analyzed (Participants) | 151 | 142
Participants | 4 | 14

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected through 30 days post-transplant or initial hospital discharge. Liver-graft related serious adverse events (LGRSAEs) were collected through 6 months post-transplant, and ischemic biliary complications were collected through 12 months post-transplant. All-cause mortality is reported through 12-months post transplant.
Description: Only death and serious adverse events were assessed. All-Cause Mortality was assessed in 153 participants in the "OCS Liver System" Arm and 147 participants in the "Control" Arm. Serious Adverse Events were monitored in 153 participants in the "OCS Liver System" Arm and 146 participants in the "Control" Arm.
Arm/Group | OCS Liver System | Control
All-Cause Mortality (participants affected / at risk) | 9/153 | 10/147
Serious Adverse Events (participants affected / at risk) | 82/153 | 72/146
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS Liver System (N=153) | Control (N=146)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 3 (3) | 4 (4)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 2 (3)
Myocardial ischaemia (Infections and infestations) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (3)
Coeliac artery compression syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Intravascular haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 4 (4)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary ischaemia (Hepatobiliary disorders) | 4 (4) | 14 (14)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic artery stenosis (Hepatobiliary disorders) | 2 (2) | 4 (4)
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein occlusion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 5 (5) | 7 (8)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal peritonitis (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 3 (3) | 0 (0)
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 13 (13) | 6 (6)
Drug toxicity (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 4 (4) | 11 (11)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 5 (5) | 7 (7)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Liver function test abnormal (Investigations) | 2 (2) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (2)
Convulsion (Nervous system disorders) | 2 (2) | 5 (5)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 4 (4)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 11 (11) | 7 (7)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Reexpansion pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Incisional drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Air embolism (Vascular disorders) | 0 (0) | 1 (1)
Artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Reperfusion injury (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Vascular shunt (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT02522871/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT02522871/SAP_001.pdf